CLINICAL TRIAL: NCT04858698
Title: Reduction Or Elimination Of Radiation During Implantation of Cardiac Devices Using Ultrasound (RADICAl USe)
Brief Title: Reduction Or Elimination Of Radiation During Implantation of Cardiac Devices Using Ultrasound
Acronym: RADICAL USE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Habib Khan (Other)
Responsible Party: Sponsor-Investigator, Habib Khan, Assistant Professor in Cardiology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10510
Record Dates: First submitted 2021-04-08; First posted 2021-04-26 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Bradycardia; Brady-tachy Syndrome
MeSH Terms: conditions — Bradycardia | interventions — Ultrasonography; Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced fluoroscopy arm (Experimental): Patients exposed to 20 seconds or less of fluoroscopy to implant a single chamber device with aid of ultrasound / echocardiography.
  Interventions: Device: Ultrasound / Echocardiography
- Conventional arm (Active Comparator): Patients exposed to more than 20 seconds of fluoroscopy to implant a single chamber device with/without the aid of ultrasound / echocardiography.
  Interventions: Device: Ultrasound / Echocardiography

INTERVENTIONS:
Device: Ultrasound / Echocardiography — Ultrasound will be used to guide vascular access and to place a lead into the right ventricle.
  Other Names: Echocardiography by using St Jude - Zonaire ultrasound and P4-1c transducer.

SUMMARY:
Specialized equipment is required to put pacemakers in the heart. This requires use of radiation to see the wires or leads being implanted in the heart. Repeated radiation use can result in permanent injury to the patient and to the doctor. The investigators aim to investigate if they can use ultrasound to guide and help in the implantation of leads into the heart. Ultrasound is a safe method and requires only a small handheld probe and a small screen to see different structures in the heart. If ultrasounds proves successful as a tool to reduce radiation then this would be very useful technical breakthrough. It would help develop smaller centres where pacemakers can be implanted without purchasing xray equipment and expensive setups.

DETAILED DESCRIPTION:
Radiation quantity used in medicine is expanding year on year with increasing clinical uses for medical illnesses and to visualize instruments being used during procedures such as cardiac devices including pacemakers. The effects of radiation are not only on the patients for their procedure but also a cumulative effect of radiation on the operators. The stochastic effects of radiation have been well reported in the literature. Advancing technologies such as 3-dimensional(3D) mapping systems have allowed for leads to be identified using a 3D matrix and safely deployed to the myocardium. However, there are significant costs associated with the use of 3D mapping systems resulting in this approach not being widely adopted. Ultrasound use during implantation of cardiac implantable electronic devices (CIED) has been utilized in the past to gain vascular access via the axillary vein with good safety results. Experimental studies to visualize leads in the heart and venous systems using 3D ultrasound showed optimism but has not translated to clinical use due to lack of technology to improve the spatial and temporal resolution. The technology in imaging resolution has improved over the last 5 years and likely can be used to visualize a pacing lead in the heart. Techniques such as intravascular cardiac ultrasound have been used to assist in implanting lead via coronary sinus in individuals who can have contrast allergies. Therefore, transthoracic echocardiogram and ultrasound should be now of sufficient quality to allow for successful pacemaker insertion.

To date, there has not been a feasibility study to evaluate complete ultrasound and echocardiography-assisted pacemaker insertion.

In this study, the investigators aim to utilize ultrasound and echocardiography to gain vascular access and to direct the pacing lead into the right ventricle to allow for safe pacemaker implantation. If this is successful, then this will allow for a larger study to be conducted for single chamber devices including implantable cardioverter defibrillators. Moreover, the investigators will be able to analyze the cost-effectiveness of this new technique compared to the conventional technique of pacemaker implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old.
2. Suitable to have either a single chamber pacemaker or single chamber cardioverter-defibrillator.

Exclusion Criteria:

1. BMI >30.
2. Pregnancy.
3. Implantation of dual-chamber and CRT devices.
4. Claustrophobia.
5. Tender chest wall or history of trauma to the chest wall.
6. Higher signal interference using ultrasound due to the presence of other medical devices or tools used in previous surgical procedures such as sternal wires, mechanical valves, breast implants.
7. History of radiation to the chest wall for oncology treatments.
8. Active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Success of implanting a single chamber lead with use of ultrasound | 0 day
  Binary outcome - successful or not.

SECONDARY OUTCOMES:
Duration of radiation will be measured in seconds | during procedure
  Comparison between the treatment and control group
Total radiation dose will be collected in centiGray and milliGray units. | during procedure
  Comparison between the treatment and control group

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre Res. Inc. (Ont.), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan HR, Triemstra S, Pardo A, Moustafa AT, Mokhtar AT, Antiperovitch P, Saravu S, Mtwesi V, Gula LJ, Leong-Sit P, Manlucu J, Yee R, Tang A. Fluoroless Implantation of Pacemaker and Cardioverter-Defibrillator Using Ultrasound As An Imaging Tool: A Multi-Operator Experience in Radical Use Study. Can J Cardiol. 2025 Dec 23:S0828-282X(25)01596-X. doi: 10.1016/j.cjca.2025.11.052. Online ahead of print. PMID 41448266